CLINICAL TRIAL: NCT02065232
Title: A Randomized, Double-blinded, Controlled Clinical Trial Comparing Post-injection Site Pain of Technetium-labeled Tilmanocept Versus Technetium-labeled Sulfur Colloid in Patients Undergoing Sentinel Lymph Node Mapping Procedure for Breast Cancer
Brief Title: Sentinel Lymph Node Mapping Post-Injection Site Pain
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SLNPain01
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tilmanocept: Patients will receive technetium-labeled tilmanocept, which is FDA approved for sentinel lymph node mapping in breast cancer.
  Interventions: Drug: Tilmanocept
- Sulfur Colloid: Patients will receive technetium-labeled sulfur colloid, which is FDA approved for sentinel lymph node mapping in breast cancer.
  Interventions: Drug: Sulfur Colloid

INTERVENTIONS:
Drug: Tilmanocept
  Other Names: Lymphoseek
  Groups: Tilmanocept
Drug: Sulfur Colloid
  Groups: Sulfur Colloid

SUMMARY:
This is a pain survey study that will compare the level of discomfort experienced by breast cancer patients after injection of either technetium-labeled sulfur colloid or technetium-labeled tilmanocept, both FDA-approved agents used for sentinel lymph node biopsy (SLNB). Breast cancer patients who are already scheduled for SLNB as part of their original surgical plan will be asked to participate in this study and be randomized to receive either technetium-labeled sulfur colloid or technetium-labeled tilmanocept. After injection, patients will complete pain questionnaires to measure the amount of discomfort they are feeling during and after they receive the injection. There will be no change to the patient's treatment plan other than the addition of pain questionnaires. The investigators' hypothesis is that patients will feel less discomfort after injection of tilmanocept versus sulfur colloid.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of biopsy-proven primary breast cancer or a diagnosis of pure ductal carcinoma in situ (DCIS) who will be undergoing intraoperative lymphatic mapping as part of their standard surgical plan.
* The patient has provided written informed consent before participating in the study, as has his/her responsible caregiver, if applicable.
* The patient is a candidate for surgical intervention, with lymph node mapping being a part of the surgical plan.
* The patient is greater than 18 years of age at the time of consent.
* The patient has an performance status of Grade 0 - 2.
* The patient has a clinical negative node status at the time of study entry.
* If the patients is of child bearing potential, the patient has a negative pregnancy test within 72 hours prior to administration of radiopharmaceutical, has been surgically sterilized, or has been postmenopausal for at least 1 year.

Exclusion Criteria:

* The patient is pregnant or lactating.
* The patient has clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients, aged 18 years or older with a diagnosis of primary breast cancer or ductal carcinoma in situ (DCIS) with planned Sentinel node biopsy (SLN) biopsy as part of the surgical plan were approached at preoperative clinic visits of the principal investigator. (Anne Wallace)
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline level of discomfort | 1,2,3,4,5,15, 30 minutes after injection
  After injection of either tilmanocept or sulfur colloid, patients will be asked to fill out a pain questionnaire at the above time points.

SECONDARY OUTCOMES:
Visualization of Sentinel Lymph Nodes on Lymphoscintigraphy | 15,30,60 minutes after injection
  After injection of sulfur colloid or tilmanocept, patients will undergo lymphoscintigraphy imaging (as is standard of care for sentinel lymph node mapping) at 5, 30, and 60 minutes. We will analyze the time it takes for sentinel lymph nodes to appear on these images comparing tilmanocept versus sulfur colloid.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States